CLINICAL TRIAL: NCT05815927
Title: Pembrolizumab and Radiotherapy for OLigometastatic Squamous Cell Carcinoma of the Head and Neck: a Randomized Phase III Study
Brief Title: Pembrolizumab and Radiotherapy for Oligometastatic Head and Neck Cancer
Acronym: PROLoNg
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Swiss Cancer Institute (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2014-HNCG; 2023-504478-39-00 (Other: EU trial number)
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Squamous Cell Carcinoma of the Head and Neck
Keywords: Pembrolizumab; Stereotactic ablative radiotherapy; oligometastatic HNSCC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : Standard of Care (Active Comparator): Pembrolizumab at a dose of 400mg every 6-weeks (Q6W) for a duration of 2 years (i.e 17 cycles) as per Standard of Care treatment of oligometastatic HNSCC disease. Palliative radiotherapy to oligometastatic disease is allowed if necessary as per standard of care to relieve symptomatic disease and prevent complications. Recommended dose regimens are 1x 8 Gy, 5x 4 Gy and 10x 3 Gy. Planning technique and target volume definition should be according to institutional standards.No ablative-stereotactic dose and no boost techniques are allowed with the exception of CNS-metastases treatment.
  Interventions: Drug: Pembrolizumab
- Arm 2 : Standard of Care + stereotattic ablative radiation (SABR) (Experimental): The Experiemnt Arm consists of pembrolizumab at a dose of 400mg every 6-weeks (Q6W) for a duration of 2 years (i.e 17 cycles) as per Standard of Care treatment of oligometastatic HNSCC disease in combination with SABR. For each oligometastatic lesion treatment, specific SABR fractions and targeted dose(Gy) should be used depending on the location of the lesion. Three-fraction regimens will deliver a fraction every second day, and five-fraction regimens are delivered daily. All treatments have to be completed within 10 working days.
  Interventions: Drug: Pembrolizumab; Radiation: stereotattic ablation radiotherapy (SABR)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab: 400mg Q6W up to 2 years (i.e 17 cycles).
Radiation: stereotattic ablation radiotherapy (SABR) — Total dose and number of fractions will depend on the site of the disease. Three-fraction regimens will deliver a fraction every second day, and five-fraction regimens are delivered daily. All treatments have to be completed within 10 working days.
  Other Names: SBRT
  Arms: Arm 2 : Standard of Care + stereotattic ablative radiation (SABR)

SUMMARY:
This is a randomized open-label multicentre phase III superiority study of the effect of adding SABR to the standard of care treatment pembrolizumab on progression free survival in patients with oligometastases of a squamous cell carcinoma of the head and neck (SCCHN), histological confirmation of the primary disease at first diagnosis, and PD-L1 CPS ≥1. After eligibility check and signing informed consent, all patients will be prospectively enrolled in a 1:1 ratio between current standard of care treatment (pembrolizumab, Arm 1) vs. SABR + standard of care treatment (Arm 2) to oligometastases.

Any radical treatment to the synchronous primary/ recurrent primary tumor and/or involved cervical nodes (surgery or radiotherapy), as decided by the local tumor board/ treating physicians, should be completed prior to enrolment.Surgical removal of metastases is allowed for diagnostic purposes or for brain metastases, as long as these metastases count toward the total number of 5 and at least one metastasis is left for treatment with SABR. Such surgical procedures should be performed prior to enrolment.

ELIGIBILITY:
Main inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent
* Histologically confirmed HNSCC of the oral cavity, oropharynx, hypopharynx, larynx or cervical primary occult and histologically or radiologically confirmed oligometastatic disease. Histological characterization of one metastatic lesion is strongly recommended.
* Patients with synchronous or metachronous oligometastatic disease according to the ESTRO/EORTC consensus (1-5 metastatic lesions, with or without primary/recurrent primary tumour and/or regional disease).
* Amenable to first-line systemic treatment for R/M SCCHN.
* For patients with oropharyngeal cancer: HPV status using p16 IHC evaluated locally.
* PD-L1 CPS of at least 1 as evaluated locally.
* Staging not older than 12 weeks before enrolment.
* All the 1-5 metastases must be amenable to SABR.
* Eligible for treatment with pembrolizumab.
* Have measurable disease based on RECIST 1.1.
* ECOG performance status of 0 to 1.
* Participants must have recovered from all treatment-related toxicities to baseline or grade ≤1, such as from previous radiotherapy, systemic treatment or surgery, and not requiring corticosteroids for managing treatment-related side effects.
* Adequate Organ Function Laboratory Values.
* Before patient registration/enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations.

Main exclusion Criteria:

* Nasopharynx, sino-nasal, and salivary gland cancers are excluded.
* In-field progression in < 6 months after curative intended locoregional irradiation of the head and neck.
* Lesions larger than 6 cm in the largest dimension as measured in the diagnostic CT or MRI scan for lesions outside the brain. Note: bone metastases over 6 cm may be included if in the opinion of the local radiation oncologist they can be treated safely and no inner organ is affected.
* Brain metastases only.
* Has received any previous radiotherapy to any of the 1-5 metastases that would be subject to SABR in the experimental arm unless the investigator agrees to treat only after discussion with the RTQA team.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Previously treated brain metastases that are radiologically non-stable. Patients with previously treated brain metastases, i.e., without evidence of progression for at least 4 weeks by repeat imaging, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention, can participate.
* Known contraindication to imaging tracer or any product of contrast media and MRI contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival by RECIST 1.1 | 2.6 years after first patient in
  To assess whether SABR added to pembrolizumab improves progression-free survival in patients with HNSCC disease, PD-L1 CPS ≥1 and 1-5 metastatic lesions, as compared to pembrolizumab alone.

SECONDARY OUTCOMES:
Overall survival | 5.2 years after first patient in
  To assess whether SABR added to pembrolizumab improves OS
Disease-specific survival | 5.2 years after first patient in
  To assess whether SABR added to pembrolizumab improves disease-specific survival
Time to disease progression | 5.2 years after first patient in
  To assess whether SABR added to pembrolizumab improves time to disease progression
Time to development of new metastatic lesions | 5.2 years after first patient in
  To assess whether SABR added to pembrolizumab improves time to development of new metastatic lesions
Time to progression in oligometastatic lesions initially present at enrolment | 5.2 years after first patient in
  To assess whether SABR added to pembrolizumab improves time to progression in oligometastatic lesions initially present at enrolment
Adverse events according to CTCAE version 5.0 | 5.2 years after first patient in
  To evaluate the safety and tolerability according to CTCAE v5.0 of SABR combined with pembrolizumab
Health-related quality of life evaluated using self-administered EORTC QLQ-C30 questionnaire | 5.2 years after first patient in
Health-related quality of life evaluated using self-administered EORTC QLQ-HN43 questionnaire | 5.2 years after first patient in
Health-related quality of life evaluated using self-administered EORTC IL-198 questionnaire | 5.2 years after first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Belermpas, MD, Study Chair — University of Zurich; Jean-Pascal Machiels, MD, Study Chair — Clinicque Universitarie Saint Luc
Locations (26):
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - CHU-UCL Namur - CHU Site Sainte-Elisabeth-UCL Namur, Namur
  - VITAZ St Niklaas - VITAZ- Oncology, Sint-Niklaas
  - Ziekenhuis aan de Stroom (ZAS) - ZAS Augustinus (previous GZA), Wilrijk
- Italy (9):
  - IRCCS--Ospedale Bellaria-Bologna, Bologna
  - AUSL - Ospedale Infermi, Faenza
  - Univ. of Florence -Azienda Ospedaliero-Universitaria Careggi, Florence
  - AUSL -Ospedale Umberto I, Lugo
  - Istituto Clinico Humanitas, Milan
  - IRCCS - Fondazione Istituto Nazionale dei Tumori, Milan
  - Azienda Sanitaria Locale Napoli 1 Centro, Napoli
  - AUSL Romagna - AUSL Della Romagna -Ospedale Santa Maria delle Croci, Ravenna
  - Azienda ospedaliero Univ Policlinico Umberto I, Rome
- Spain (5):
  - Hospital Universitari Vall d'Hebron -Vall d'Hebron Institut Oncologia, Barcelona
  - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
- Switzerland (7):
  - Kantonsspital Aarau, Aarau
  - Oncology Institute of Southern Switzerland (IOSI) - Oncology Institute of Southern Switzerland - Ospedale San Giovanni, Bellinzona
  - Inselspital - Inselspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zurich, Zurich